CLINICAL TRIAL: NCT01814475
Title: Prospective, Phase II Randomized Study to Compare Busulfan-fludarabine Reduced-intensity Conditioning (RIC) With Thiotepa-fludarabine RIC Regimen Prior to Allogeneic Transplantation of Hematopoietic Cells for the Treatment of Myelofibrosis
Brief Title: Study to Compare Busulfan-fludarabine With Thiotepa-fludarabine Regimen in Allogeneic Transplantation for Myelofibrosis
Acronym: GITMO-MF2010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-022052-23 GITMO - MF2010
Record Dates: First submitted 2013-03-14; First posted 2013-03-20 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Myelofibrosis
Keywords: myelofibrosis; unfavourable prognostic factors; Allogeneic stem cell transplantation; Progression Free Survival; thrombocythemia vera; polycythemia vera; Reduced-intensity conditioning
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — Busulfan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Fludarabine + Busulphan (Active Comparator): Conventional conditioning regimen with Fludarabine and Busulphan (Busilvex)for allogeneic stem cell transplantation in myelofibrosis
  Interventions: Drug: A: Fludarabine + Busulphan
- B: Fludarabine + Thiotepa (Experimental): Reduced-intensity conditioning with Fludarabine and Thiotepa for allogeneic stem cell transplantation in myelofibrosis
  Interventions: Drug: B: Fludarabine + Thiotepa

INTERVENTIONS:
Drug: A: Fludarabine + Busulphan — Fludarabine 30 mg/m2/d, day -8 to day-3 and Busulphan (Busilvex) 0,8 mg/Kg/i.v. dose x 4 doses on days -5,-4 and x 2 doses on day -3, total dose 8 mg/Kg) prior allogenic transplant (day zero)
  Other Names: BU-FLU
  Arms: A: Fludarabine + Busulphan
Drug: B: Fludarabine + Thiotepa — Fludarabine 30 mg/m2/d day -8 to day -3 Thiotepa 6 mg/Kg for 2 doses ( days -4, -3) prior allogeneic transplant (day zero)
  Other Names: THIO-FLU
  Arms: B: Fludarabine + Thiotepa

SUMMARY:
This study will be performed as a prospective multicenter phase II trial for compare busulfan-fludarabine reduced-intensity conditioning (RIC) with thiotepa-fludarabine RIC regimen prior to allogeneic transplantation of hematopoietic cells for the treatment of myelofibrosis.

The primary endpoint for this study is to compare Progression Free Survival of two different RIC regimens for allogeneic stem cell transplantation in myelofibrosis.

Progression Free Survival is defined as the time from the date of randomization to the date of the first documented disease progression or relapse (according to the International Working Group Consensus Criteria) or death due to any cause. Patients who have neither progressed nor died at the time of study completion or who are lost to follow-up are censored at the data of the last follow up for progression of disease for this study.

DETAILED DESCRIPTION:
This is the first study to explore the efficacy of two different Reduced-intensity conditioning (RIC) regimens for allogeneic stem cell transplantation in myelofibrosis. The choice of 60 patients is based on feasibility reasons. GITMO data at hand points to an estimated accrual of twenty patients per year over a tree-year enrolment period. Criteria for defining sample size do not follow statistical power estimates in order to demonstrate the difference of lack of it between two treatments. However, the criteria reflect the overall efficacy and safety of comparing the two treatments among all patients requiring the treatment within the health system. This criterion offers the best estimate for power of study.

Myelofibrosis is a clonal hematopoietic stem cell disorder that is clinically characterized by progressive anemia, marked splenomegaly, extramedullary hematopoiesis, constitutional symptoms and a significant risk of evolution into acute leukaemia myelofibrosis can appear as a primitive or idiopathic disorder or, less frequently, as a secondary complication of essential thrombocythemia or polycythemia vera, with a clinical presentation and course similar to the idiopathic form. The disease affects mainly elderly people, with a median age at diagnosis of about 65 years. It is a heterogeneous disorder in term of presentation and evolution, with a median overall survival (OS) varying between 2 and 15 years, depending on the presence or absence of clinically defined prognostic factors. Adverse prognostic factors for survival have included advanced age, marked anemia, leukocytosis or leukopenia, abnormal karyotype, constitutional symptoms and presence of circulating blasts. Moreover, the prognostic value of cytogenetic abnormalities, increased number of circulating cluster of differentiation 34 cells in peripheral blood and Janus kinase 2 mutational status has been also evaluated. The available prognostic score systems are mainly based on clinical variables. The most widely used is the 'Lille score' (Dupriez et al.) which is based on hemoglobin level and leukocyte count. The Mayo Clinic Group tried to improve the Lille score by adding thrombocytopenia and monocytosis. The International Working Group for Myelofibrosis Research and Treatment recently proposed a new scoring system analyzing the largest patient population and recognized 5 main unfavourable variables which were: age > 65 years, presence of constitutional symptoms, and circulating blasts cells ≥ 1%, anemia and leucocytosis. All these prognostic systems could clearly separate intermediate or high risk patients (with a median survival ranging between 1 and 4 years) from patients with a favourable prognosis (median survival of 8-10 years).

Kroger on behalf of the European Group for Blood and Marrow Transplantation reported data on 104 patients mainly with intermediate or high risk score who received a conditioning regimen based on fludarabine 180 mg/mq and busulfan 8 mg/kg i.v or 10 mg/Kg p.o and hematopoietic stem cells coming from sibling or unrelated donors. Engraftment was 99%; 1-year transplant-related mortality was 16% and was significantly increased in patients older than 50 years, in cases with intermediate and high-risk myelofibrosis and after transplants from mismatched donors. Five-year overall survival was 67% and 5 -year event-free-survival was 51%. Relapse rate was higher in splenectomized patients and if disease duration prior transplant was >24 months. Moreover, Kroger reported that this conditioning regimen induced a Janus kinase 2 negativity in 78% of patients carrying the V617-JAK2 mutation before transplant and produced a rapid regression of bone marrow fibrosis in 59% of patients al day +100 and in 100% of patients at day +360. At present, the busulfan-fludarabine regimen could be considered as the Reduced-intensity conditioning regimen that has been tested on the largest patient population and demonstrated the best results in terms of feasibility and clinical, molecular and histological responses.

The Principal Investigator has recently reported data on a population of 100 patients with myelofibrosis who underwent allogeneic hematopoietic stem cell transplantation in 26 transplant centers that are part of the GITMO in a 20-year period between 1986 and 2006 and we retrospectively analyzed the influence of patient and disease clinical features before stem cell transplantation and of transplant procedures on transplant-related mortality (TRM) and overall survival. We confirmed that myelofibrosis remains a rare indication for stem cell transplantation with the recruitment of about 15-17 cases per year since 2002 and observed a great heterogeneity in terms of conditioning regimens, Graft versus Host Disease prophylaxis and supportive measures. Although we observed a significative and progressive improvement of transplant-related mortality after 1996, we couldn't recognized any significative difference in outcome either between patients treated with myeloablative versus reduced- intensity regimens or among those treated with different Reduced-intensity conditioning regimen. The lack of any association between intensity of conditioning or type of drugs included in the preparative regimen could be in part due to the great heterogeneity of transplant procedures. However, we showed that the regimens including thiotepa were administered to 24 out 52 patients (46%), whereas the other patients received heterogeneous preparative regimens. The combination of thiotepa and cyclophosphamide was originally described for autologous transplants; then thiotepa was used with a 30% dose reduction as Reduced-intensity conditioning regimen in association with Cyclophosphamide and/or fludarabine followed by haematopoietic stem cells in elderly patients with acute leukemias, in heavily pretreated relapsed or refractory lymphomas and in myelodysplastic syndromes, showing to be highly feasible and effective. Both these protocols were used in Italy by researchers and physicians participating to GITMO.

In conclusion, the rational of the present study are the following:

* myelofibrosis is a rare indication for allogeneic transplantation with a limited number of patients recruitable in the whole Italian region.
* At the present time there are not available sufficient data to support a standard conditioning regimen for these patients.
* Italian hematologists grouped in the GITMO intend to overcome the general uncertainty in the choice of the conditioning regimen and to test prospectively in a controlled study a uniform strategy of transplant procedures for this rare condition.
* Therefore, we want to compare two Reduced-intensity conditioning regimens, the thiotepa-fludarabine regimen, that has been the most common one used in Italy in the last 5 years , and the busulfan-fludarabine one, that has been reported in the literature to achieve the best results in terms of feasibility and clinical responses . A randomized comparison is likely to increase our knowledge on safety and efficacy of these conditioning regimens and consolidate assumption for the planning of a phase II trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ≤ 70 years
* Primary or secondary myelofibrosis after essential thrombocythemia or polycythemia vera
* One of the following unfavourable prognostic factors: Hb < 10 g/dL or leukocytes >25x109/L or > 1% circulating blasts in the peripheral blood or constitutional symptoms
* Performance Status (Karnofsky)≥ 60%
* Hematopoietic Cell Transplantation Comorbidity Score ≤ 5
* Written informed consent

Exclusion Criteria:

-≥ 20% blasts in peripheral blood and/or bone marrow

* Positive serologic markers for human immunodeficiency virus (HIV)
* Acute hepatitis B virus (HBV) or acute hepatic C virus (HCV) infection
* Severe irreversible renal, hepatic, pulmonary or cardiac disease, such as: --total bilirubin, Serum Glutamate Oxaloacetate Transaminase (SGOT) or Serum Glutamate Pyruvate Transaminase (SGPT) > 5 the upper normal limit;

  * Left ventricular ejection fraction < 40%;
  * Clearance creatinine < 30 ml/min;
  * Diffusing Capacity of Lung for Carbon monoxide (DLCO) < 30% and/or receiving supplementary oxygen.
* Pregnancy or lactation
* Any active, uncontrolled infection

Donors:

* Age ≥ 18 < 65 years
* human leukocyte antigen (HLA)-identical sibling donor by high resolution DNA-based HLA-A, -B, -C, -DRB1, typing
* human leukocyte antigen (HLA)-identical unrelated donor by high resolution DNA-based human leukocyte antigen-A, human leukocyte antigen-B, human leukocyte antigen-C, human leukocyte antigen-DRB1 typing. One allele mismatched (class I) can be accepted for recipients up to 60 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-07; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Progression -free survival at one year | Assessment at 1 year post randomization
  The primary endpoint for this study is to compare Progression Free Survival of two different RIC regimens for allogeneic stem cell transplantation in myelofibrosis.
  Progression Free Survival is defined as the time from the date of randomization to the date of the first documented disease progression or relapse (according to the International Working Group Consensus Criteria) or death due to any cause. Patients who have neither progressed nor died at the time of study completion or who are lost to follow-up are censored at the data of the last follow up for progression of disease for this study.

SECONDARY OUTCOMES:
Safety and efficacy profile: The non relapse mortality | Assessment at 1 year post randomization
  The non relapse mortality (NRM) is defined as death due to any other cause than progression of malignancy after allogeneic stem cell transplantation.
Safety and efficacy profile: Overall survival | Assessment at 1 year post randomization
  Overall survival is defined as the time between randomization and the date of death due to any cause or the last date the patient was known to be alive (censored observation) at the date of the data cut-off for the final analysis
Safety and efficacy profile: responses | Assessment at 1 year post randomization
  Rate of clinical hematological and histological responses
Safety and efficacy profile: molecular remissions | Assessment at 1 year post randomization
  Rate of molecular remissions in patients having a molecular marker (according to IWG consensus criteria)
Safety and efficacy profile: engraftment | participants will be followed for the duration of hospital stay, an expected average of 30 days
  Cumulative incidence of engraftment. The day of engraftment is defined as the first 3 consecutive days on which the blood granulocyte count rises to 0.5 x 109/L
Acute Graft-versus-Host Disease (aGvHD) | from date of transplant to until the date of first event of aCGVD assessed up to 100 days post transplant
  The available information in the European Group for Blood and Marrow Transplantation (EBMT) data regard the date of onset and the maximum grade of aGvHD. It is therefore possible to estimate the probability of aGvHD in a competing risks setting (death is a competing event; whether relapse/progression is a competing event must be discussed with the physician). By definition, patients alive (relapse/progression-free) at day 100 without having experienced aGvHD are censored. If the dates of onset are missing for the majority of patients, the analysis can focus only on the occurrence of aGvHD, which is analyzed by a logistic regression model. This method would however be incorrect if there is a (non negligible) percentage of censored observations or if competing events occurred before day 100.
Chronic Graft-versus-Host Disease (cGvHD) | from day +100 post transplant to until the date of first event to cGVHD assessed up to 1 years post enrolment
  When possible, if information on the date of 1°occurrence of cGvHD is available, it should be analyzed as a time-to-event outcome, being death (and possibly relapse/progression) the competing event; data are censored for patients alive (relapse/progression-free) without episodes of cGvHD at last follow-up. Since cGvHD is defined only for patients surviving at least 100 days, the survival model should consider a left truncation at 100 days; alternatively, the time of occurrence of cGvHD must be computed from 100 days. If information on the timing of cGvHD is not available, the outcome considered is the occurrence, and the statistical model to be used is the logistic regression. Only patients surviving at least 100 days are considered to be at risk of developing cGvHD, therefore the analysis must be restricted to these patients. This analysis is of course not satisfactory because it does not take into account the occurrence of death and censoring.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Patriarca, MD, Principal Investigator — Azienda Ospedaliera Santa Maria della Misericordia di Udine
Locations (21):
- Italy (21):
  - Azienda Ospedaliera SS Antonio e Biagio, Alessandria
  - Clinica di Ematologia - Ospedali Riuniti di Ancona, Ancona
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - Ospedale Ferrarotto - Ematologia, Catania
  - Cattedra di Ematologia - Azienda Ospedaliera di Careggi, Florence
  - Ematologia e Centro Trapianti Midollo Osseo - Ospedale IRCCS Casa Sollievo della Sofferenza, Foggia
  - AOU IRCCS San Martino - IST, Genova
  - Ospedale Panico, Lecce
  - Divisione di Ematologia - Istituto Nazionale dei Tumori, Milan
  - Divisione Ematologia - Azienda Ospedaliera Universitaria - Policlinico -, Modena
  - AO Ospedali Riuniti Villa Sofia - Cervello, Palermo
  - Dipartimento Oncologico La Maddalena, Palermo
  - Fondazione IRCCS San Matteo, Pavia
  - Dip. di Ematologia - Unità di Terapia Intensiva Ematologica per il Trapianto Emopoietico - Ospedale Civile di Pescara, Pescara
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - Arciospedale S. M. Novella, Reggio Emilia
  - Cattedra di Ematologia - Università La Sapienza, Roma
  - Ospedale San Giuseppe Moscato, Taranto
  - Ematologia 2 - ASO San Giovanni Battista, Torino
  - A.O. Santa Maria della Misericordia, Udine